CLINICAL TRIAL: NCT06536244
Title: Impact of Perioperative Anesthetic Management on Renal Cancer Progression.
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0380
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Perioperative Anesthetic; Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The relationship between perioperative drugs, including preoperative medications, anesthetics, and analgesics, and postoperative outcomes in cancer patients is a complex and evolving field of study. Understanding how those medications might impact outcomes such as pain, acute kidney injury, and recurrence is crucial for optimizing perioperative care in renal cancer patients.

DETAILED DESCRIPTION:
This retrospective study will investigate the association of perioperative drugs on short and long-term postoperative outcomes in patients undergoing kidney surgeries for renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Participants (18 years of age or older)
2. Participants having radical or partial nephrectomies with curative intent.

Exclusion Criteria:

1. Patients with distant metastatic disease and those with multiple (more than 1) primary tumors at the time of the nephrectomy
2. Biopsies
3. Participants who had radiofrequency or microwave ablations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 72 hours and 30 days postoperatively

SECONDARY OUTCOMES:
Overall survival | Recurrence-free survival:The length of time from surgery to last seen without recurrence or with recurrent disease.
  The length of time from surgery to last follow-up alive or death.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org